CLINICAL TRIAL: NCT01367093
Title: French and EuRopean Outcome Registry in Intensive Care Unit
Acronym: FROG-ICU
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI10029; 2010-A01374-35 (Other: IDRCB)
Record Dates: First submitted 2011-05-27; First posted 2011-06-06 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-04

CONDITIONS: Intensive Care Unit Syndrome; Tracheal Intubation Morbidity
Keywords: BIOLOGICAL MARKERS; INTENSIVE CARE UNIT; MORTALITY; QUALITY OF LIFE; CARDIOVASCULAR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and urine at admission and ICU discharge
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU patients admitted for severe illness

SUMMARY:
The purpose of this study is to identify within a cohort of ICU patients admitted for severe illness those who are at risk of death in the year following the discharge from ICU.

DETAILED DESCRIPTION:
FROG-ICU is an epidemiological, observational, prospective, multi centric, cohort study designed for description, prognostic and evaluation. This trial includes as a first step a complete registry of patients admitted to the ICU and as a second step, the outcome of the patients at 1 year after they have been discharged alive from ICU.

Plasma and urine samples will be with drawn biomarkers measurements at admission and ICU discharge. It is a multicentric study involving 1 center in Belgium et 24 centers in France.

ELIGIBILITY:
Inclusion criteria:

* Adult patients hospitalized in ICU
* Patients should have been intubated more than 24 hours
* or treated with a positive inotropic agent for more than 24 hours (if not ventilated

Exclusion Criteria:

* age < 18 years
* pregnancy women
* Breast-feeding women
* Not affiliated with social security
* Dying man
* End of life patient
* Traumatic Brain Injury (IGCS < 8)
* NTBR
* vegetative coma
* Transplanted for less than year
* no french speaking patient
* out of france resident
* end of life decision during the following

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients admitted for severe illness those who are at risk of death in the year following the discharge from ICU.
Sampling Method: Probability Sample
Enrollment: 2137 (Actual)
Dates: Start 2011-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
All cause mortality at one year after ICU discharge | one year

SECONDARY OUTCOMES:
To assess quality of life in the year following a stay in ICU | one year
To identify key determinants of cardiovascular morbidity and mortality in the year following a stay in ICU | one year
To investigate the performance of plasma biomarkers usually measured in ICU, to assess the risk of death during the stay in ICU and one year after the discharge. | one year
To set up a biological collection of plasma and urine, in order to measure new plasma biomarkers in the assessment of prognosis in the year following a stay in ICU. | one year
to evaluate social conditions | one year

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Mebazaa, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Department of Anesthesiology and Intensive Care Unit - Lariboisiere Hospital, Paris
  - St Louis hospital, department of intensive care, Paris

REFERENCES:
- [Result] Mebazaa A, Casadio MC, Azoulay E, Guidet B, Jaber S, Levy B, Payen D, Vicaut E, Resche-Rigon M, Gayat E. Post-ICU discharge and outcome: rationale and methods of the The French and euRopean Outcome reGistry in Intensive Care Units (FROG-ICU) observational study. BMC Anesthesiol. 2015 Oct 12;15:143. doi: 10.1186/s12871-015-0129-2. PMID 26459405
- [Derived] Blet A, Walter-Petrich A, Cherifa M, Bruno J, Tran Dinh A, Azoulay E, Chousterman B, Cotter G, Davison B, Deniau B, Gayat E, Guidet B, Harrois A, Kimmoun A, Leone M, Wittebole X, Ambrosy AP, Mebazaa A, Resche-Rigon M. Survival after ICU discharge is shaped more by chronic disease than admission severity. J Crit Care. 2026 Apr;92:155401. doi: 10.1016/j.jcrc.2025.155401. Epub 2025 Dec 10. PMID 41380507
- [Derived] Borouchaki A, de Roquetaillade C, Boutin L, Gayat E, Mebazaa A, Chousterman BG. Association between serum uric acid level and outcome in intensive care unit, an ancillary analysis of the FROG-ICU cohort (URIC-ICU). Anaesth Crit Care Pain Med. 2025 Nov;44(6):101610. doi: 10.1016/j.accpm.2025.101610. Epub 2025 Sep 29. PMID 41033450
- [Derived] Pharaboz A, Kimmoun A, Gunst J, Duarte K, Merkling T, Gayat E, Mebazaa A, Glenn-Chousterman B. Association between type II diabetes mellitus and 90-day mortality in a large multicenter prospectively collected cohort. A FROG ICU post-hoc study. J Crit Care. 2023 Feb;73:154195. doi: 10.1016/j.jcrc.2022.154195. Epub 2022 Oct 27. PMID 36368176
- [Derived] Blet A, McNeil JB, Josse J, Cholley B, Cinotti R, Cotter G, Dauvergne A, Davison B, Duarte K, Duranteau J, Fournier MC, Gayat E, Jaber S, Lasocki S, Merkling T, Peoc'h K, Mayer I, Sadoune M, Laterre PF, Sonneville R, Ware L, Mebazaa A, Kimmoun A. Association between in-ICU red blood cells transfusion and 1-year mortality in ICU survivors. Crit Care. 2022 Oct 7;26(1):307. doi: 10.1186/s13054-022-04171-1. PMID 36207737
- [Derived] Soussi S, Sharma D, Juni P, Lebovic G, Brochard L, Marshall JC, Lawler PR, Herridge M, Ferguson N, Del Sorbo L, Feliot E, Mebazaa A, Acton E, Kennedy JN, Xu W, Gayat E, Dos Santos CC; FROG-ICU; CCCTBG trans-trial group study for InFACT - the International Forum for Acute Care Trialists. Identifying clinical subtypes in sepsis-survivors with different one-year outcomes: a secondary latent class analysis of the FROG-ICU cohort. Crit Care. 2022 Apr 21;26(1):114. doi: 10.1186/s13054-022-03972-8. PMID 35449071
- [Derived] Takagi K, Akiyama E, Paternot A, Miro O, Charron C, Gayat E, Deye N, Cariou A, Monnet X, Jaber S, Guidet B, Damoisel C, Barthelemy R, Azoulay E, Kimmoun A, Fournier MC, Cholley B, Edwards C, Davison BA, Cotter G, Vieillard-Baron A, Mebazaa A. Early echocardiography by treating physicians and outcome in the critically ill: An ancillary study from the prospective multicenter trial FROG-ICU. J Crit Care. 2022 Jun;69:154013. doi: 10.1016/j.jcrc.2022.154013. Epub 2022 Mar 9. PMID 35278876
- [Derived] Boutin L, Legrand M, Sadoune M, Mebazaa A, Gayat E, Chadjichristos CE, Depret F. Elevated plasma Galectin-3 is associated with major adverse kidney events and death after ICU admission. Crit Care. 2022 Jan 6;26(1):13. doi: 10.1186/s13054-021-03878-x. PMID 34991653
- [Derived] Kimmoun A, Cariou A, Gayat E, Feliot E, Takagi K, Megarbane B, Mebazaa A, Deye N; FROG-ICU Study investigators. One-year outcome of patients admitted after cardiac arrest compared to other causes of ICU admission. An ancillary analysis of the observational prospective and multicentric FROG-ICU study. Resuscitation. 2020 Jan 1;146:237-246. doi: 10.1016/j.resuscitation.2019.10.021. Epub 2019 Oct 31. PMID 31678408
- [Derived] Cinotti R, Voicu S, Jaber S, Chousterman B, Paugam-Burtz C, Oueslati H, Damoisel C, Caillard A, Roquilly A, Feuillet F, Mebazaa A, Gayat E; FROG-ICU investigators. Tracheostomy and long-term mortality in ICU patients undergoing prolonged mechanical ventilation. PLoS One. 2019 Oct 2;14(10):e0220399. doi: 10.1371/journal.pone.0220399. eCollection 2019. PMID 31577804
- [Derived] Legrand M, Hollinger A, Vieillard-Baron A, Depret F, Cariou A, Deye N, Fournier MC, Jaber S, Damoisel C, Lu Q, Monnet X, Rennuit I, Darmon M, Zafrani L, Leone M, Guidet B, Friedman D, Sonneville R, Montravers P, Pili-Floury S, Lefrant JY, Duranteau J, Laterre PF, Brechot N, Oueslati H, Cholley B, Launay JM, Ishihara S, Sato N, Mebazaa A, Gayat E; French and euRopean Outcome reGistry in ICUs (FROG-ICU) Investigators. One-Year Prognosis of Kidney Injury at Discharge From the ICU: A Multicenter Observational Study. Crit Care Med. 2019 Dec;47(12):e953-e961. doi: 10.1097/CCM.0000000000004010. PMID 31567524
- [Derived] Hollinger A, Gayat E, Feliot E, Paugam-Burtz C, Fournier MC, Duranteau J, Lefrant JY, Leone M, Jaber S, Mebazaa A, Arrigo M; FROG ICU study investigators. Gender and survival of critically ill patients: results from the FROG-ICU study. Ann Intensive Care. 2019 Mar 29;9(1):43. doi: 10.1186/s13613-019-0514-y. PMID 30927096
- [Derived] Bastian K, Hollinger A, Mebazaa A, Azoulay E, Feliot E, Chevreul K, Fournier MC, Guidet B, Michel M, Montravers P, Pili-Floury S, Sonneville R, Siegemund M, Gayat E; FROG-ICU Study Investigators. Association of social deprivation with 1-year outcome of ICU survivors: results from the FROG-ICU study. Intensive Care Med. 2018 Dec;44(12):2025-2037. doi: 10.1007/s00134-018-5412-5. Epub 2018 Oct 23. PMID 30353380
- [Derived] Gayat E, Hollinger A, Cariou A, Deye N, Vieillard-Baron A, Jaber S, Chousterman BG, Lu Q, Laterre PF, Monnet X, Darmon M, Leone M, Guidet B, Sonneville R, Lefrant JY, Fournier MC, Resche-Rigon M, Mebazaa A, Legrand M; FROG-ICU investigators. Impact of angiotensin-converting enzyme inhibitors or receptor blockers on post-ICU discharge outcome in patients with acute kidney injury. Intensive Care Med. 2018 May;44(5):598-605. doi: 10.1007/s00134-018-5160-6. Epub 2018 May 15. PMID 29766216
- [Derived] Gayat E, Cariou A, Deye N, Vieillard-Baron A, Jaber S, Damoisel C, Lu Q, Monnet X, Rennuit I, Azoulay E, Leone M, Oueslati H, Guidet B, Friedman D, Tesniere A, Sonneville R, Montravers P, Pili-Floury S, Lefrant JY, Duranteau J, Laterre PF, Brechot N, Chevreul K, Michel M, Cholley B, Legrand M, Launay JM, Vicaut E, Singer M, Resche-Rigon M, Mebazaa A. Determinants of long-term outcome in ICU survivors: results from the FROG-ICU study. Crit Care. 2018 Jan 18;22(1):8. doi: 10.1186/s13054-017-1922-8. PMID 29347987
- [Derived] Legrand M, Januzzi JL Jr, Mebazaa A. Critical research on biomarkers: what's new? Intensive Care Med. 2013 Oct;39(10):1824-8. doi: 10.1007/s00134-013-3008-7. Epub 2013 Jul 5. No abstract available. PMID 23828026